CLINICAL TRIAL: NCT03964818
Title: Pressure Sore-related Osteitis Treated by Flap Coverage and Short Antibiotic Regimen
Acronym: SCAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 19ADH-SCAR
Record Dates: First submitted 2019-05-14; First posted 2019-05-28 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-05

CONDITIONS: Pressure-related Osteitis
Keywords: osteitis; flap surgery; short-course antibiotics
MeSH Terms: conditions — Osteitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pressure ulcers associated with osteitis are frequent among patients with spinal cord injury (SCI), and optimal management is not well known. In a French referral center, debridement and flap coverage surgeries performed simultaneously are followed by a short antibiotic treatment targeting the bacteria involved. The aim of the study is to evaluate patient's outcome at Day 45 after surgery, and identify factors associated with failure.

DETAILED DESCRIPTION:
Spinal cord injured (SCI) population is subject to pressure ulcers because of numerous risk factors: neurological disorders, which reduce ability to mobilization, potential, undernutrition, confinement to bed, and vascular disorders promoting the lesions.

Despite the attention given to preventative strategies, in this population, prevalence of pressure ulcers varies from 10% to 30%, with an annual incidence rates range ranging from 20%-% to 31%.

In community-dwelling SCI population, stages III and IV pressure ulcers account for 25% of total ulcers observed.

They are a major cause of healthcare centers admissions or homecare nursing. Duration of ulcers could vary from 1 week to 3 years.

Also, their occurrence is associated with potential repeated hospitalizations and with a longer length of stay. Furthermore, pressure ulcers are an important economic burden to the health care system.

Pressure ulcers interfere with the patient's physical, psychological, and social well-being and impact the overall quality of life.

Over recent years, an increased pressure ulcer prevalence has been reported. Therefore, they are frequent and their clinical spectrum is wide. They also readily become superinfected and can lead to sepsis.

Establishing the diagnosis of osteomyelitis in this setting is challenging, and physicians often struggle with the appropriate therapeutic management.

A recent review did not find evidence of benefit of antibacterial therapy in osteomyelitis associated with pressure ulcers without concomitant surgical debridement and wound coverage. But this type of management remains controversial.

In a French referral center, patients with pressure ulcer-related osteitis benefit from a one-stage surgical management with bone shaving and flap covering, followed by a probabilistic post-operative antibiotic treatment, secondarily adapted to peroperative samples, for a total duration of effective antibiotic treatment of 7 or 10 days.

Thus, the investigators aim to evaluate this original strategy, identify risk factors for failure, and focus on the role of antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years;
* Spinal cord injured patients with pressure-related osteitis treated with flap coverage and short antibiotic treatment.

Exclusion Criteria:

* Patient < 18 years;
* Patient under under guardianship;
* Patient with concomitant infections;
* Patient having declare his opposition to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal cord injured patients with pressure-related osteitis treated with flap coverage and short antibiotic treatment.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment failures at Day 45 after surgery | at 45 days
  Primary outcome is the number of patients presenting treatment failure during a 45-day follow-up period after surgery, defined as the presence of dehiscence, and/or local signs of inflammation, and/or sepsis, and/or additional antibiotic treatment.

SECONDARY OUTCOMES:
Risk factors associated with the occurrence of treatment failure at Day 45 after surgery | at 45 days
  Risk factors among patients' baseline characteristics, biological or microbiological analysis, or antibiotic treatments, significantly associated with the occurrence of treatment failure during a 45-day follow up period after surgery.
Impact of antibiotic treatment duration on the occurrence of treatment failure at Day 45 after surgery | at 45 days
  Comparison between 7 days and 10 days of antibiotic treatment duration on the number of patients presenting treatment failure at Day 45 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien DINH, MD, Principal Investigator — Infectious Diseases Department - Raymond Poincaré University Hospital
Locations (1):
- Infectious Diseases Department - Raymond Poincaré University Hospital, Garches, Hauts-de-Seine, France